CLINICAL TRIAL: NCT06461416
Title: Occupational Resilience: A Pilot Trial for a Preliminary Estimate of the Effectiveness of a Novel Theoretical Framework
Brief Title: A Trial for a Preliminary Estimate of the Effectiveness of a Novel Theoretical Framework
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 276865
Record Dates: First submitted 2024-06-10; First posted 2024-06-17 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer; Breast Cancer
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will utilize the randomized study design with two groups of 15 participants in each arm. The intervention group will receive telehealth occupational therapy services for 12 weeks. The control group will meet three times via zoom but not receive an intervention. All participants will have three assessments completed before and after the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Group A will receive telehealth occupational therapy services for 12 weeks
  Interventions: Behavioral: ActiveHeal
- Control (No Intervention): Group B will meet three times via zoom but not receive an intervention

INTERVENTIONS:
Behavioral: ActiveHeal — Participants will have 6 group activity sessions and six individualized sessions from home, all focused on optimizing persistence in performance of specific selected activities.
  Arms: Intervention

SUMMARY:
* Aim 1: To determine the preliminary effect sizes of al ActiveHeal EST (Engage-Sustain-Triumph) Program on occupational resilience.
* Aim 2: To determine the preliminary effect sizes of ActiveHeal EST (Engage-Sustain-Triumph) on health status [quality of life (QoL) and Psychological wellbeing (PWB)].
* Aim 3: To determine the extent to which ActiveHeal EST (Engage-Sustain-Triumph) Program is an acceptable and feasible Intervention for breast and prostate cancer survivors.

DETAILED DESCRIPTION:
The study will utilize the randomized study design with two groups of 15 participants each arm. The intervention group will receive occupational therapy services for 12 weeks. The control group will meet three times via zoom but not receive an intervention. All participants will have three assessments completed before and after the intervention. The experimental group will have a feasibility and acceptability survey at the end of the intervention.

Week 1-6 Recruitment, Informed Consent Process Commenced, and Randomization (Both Groups A & B) Week 7-8 Pretests: Administer Occupational Resilience Measure (ORM 1.0), World Health Organization Quality of Life Scale (WHOQOL BREF), and Psychological Wellbeing Scale. To be completed with participant via Zoom (Both Groups A & B) Week 9, 11, 15, &18 (Week 1, 2, 3, 4, 7, & 10 of the ActiveHeal EST (Engage-Sustain-Triumph)Program) Six Group ActiveHeal EST Sessions (Group A only). Each session is 75 minutes. It will include education on benefits of activity and strategies to make sustained performance possible (e.g., managing fatigue, pain, and edema), highlighting History, Experience, Benefits, and Adaptation (Location: Teams- Online). The group sessions will be led by the PI (or one of the trained occupational therapists who are familiar with the applied group and individual therapy process) and a student assistant to assist in the specified group activity performance. Although the intervention approach is specific, the use of activity as intervention is well understood by any certified occupational therapist. The training will therefore focus on what the sessions look like if these four factors are the guide to group or individual intervention, and a review of occupational therapy best practices for adults with cancer. Three additional therapists will be trained by PI in a 60 minute group session, to be able lead individual or group sessions.

Participants in the A group will receive exercise materials and handouts, a TENS unit and other resources for the individualized intervention plan. A Transcutaneous Electrical Nerve Stimulation (TENS) unit is a device that is included to help with pain control because pain often limits activity performance for cancer patients. It is not used to collect additional data but for pain control, to improve activity performance only for participants who report pain as a barrier in everyday tasks. All participants who receive the device will receive individualized education on how to use the device (during individual sessions). No information will be shared with the device manufacturer. Participants will be allowed to keep the devices to continue using it for pain control after the study. An example of an DFA-approved TENS unit is the TENS 7000 (www.tens7000.com).

ActiveHeal EST (Engage-Sustain-Triumph) group sessions will utilize a developmental group intervention model. Such intervention models allow the group to increasingly take charge of group activities and processes, with more structure and support at the beginning but members gradually take over leadership and group management roles, ideally running the group and meeting shared goals without a therapist by the end of the process . This model is selected because it has potential to enable members to develop relationships and build capacities that allow them to support one another after the intervention period. The model is also selected to allow participants to draw from benefits of group interventions, including installation of hope, universality, imparting of knowledge, altruism, corrective family re-enactment, development of socialization skills, imitative behavior, interpersonal learning, group cohesiveness, catharsis, and finding meaning.

Because these models are known to be optimal with 5-10 participants, Group A participants will be divided into two groups, but the same session plan will be used on the day of the meetings. That is, there will be two similar sessions per day of meeting, and participants will attend one session, with the same group each time. Group members will vote for their preferred activities for the upcoming meeting and the activities that are favored by the majority will be selected if consistent with group goals. These activities may include group physical exercise, healthy meal preparation activity, meditation, yoga, guided imagery, music experience (listening and/or performance) and dance.

All ActiveHeal EST (Engage-Sustain-Triumph) sessions will follow Cole's 7 steps, which are: Introduction, Activity, Sharing, Processing, Generalizing, Application, and Summary. These 7 steps will allow participants contemplate and share their experiences with a particular activity [History], demonstrate or build capacity for activity performance [Experience], reflect on health benefits of an activity [Benefits] and consider ways to sustain activity when barriers emerge []adaptation]. The 7 steps ensure that in each session group members will 1) evaluate the strategies they are using to enhance activity performance, 2) reflect or share how they have or could apply new strategies to support activity performance and health, and 3) develop an updated feasible plan of action while keeping in mind possible barriers and potential solutions to optimize activity engagement.

Each ActiveHeal EST (Engage-Sustain-Triumph) session will include a blend of 1) educational content and 2) shared activity to facilitate learning. Tentatively, the session themes include:

Optimizing lifestyle balance to improve health Psychoeducation, coping skills, relaxation Meditation/Mindfulness, yoga, creative arts Physical exercises, walking, hiking, aerobic activities Cognitive retraining Repeat of any of the above themes, based on what participants choose

Session themes about content will be retained regardless of the kind of activities selected by group members, but the sequence of themes will be determined in consultation with group members, consistent with commonly accepted group intervention guidelines.

Educational content will consistently highlight the impact of History, Experience, Benefits and Adaptation on long-term activity performance, and strategies for promoting success in enduring activity performance. Regardless of the session theme, four OR factors will be covered within Cole's last 3 steps, led by an occupational therapist and an assistant.

Week 11 & 14 (Week 3 and 6 of active study period) Control Group B Meeting via Zoom - this study meeting lasts 15 to 30 minutes allowing the PI to touch base with the control participants to see how they are doing. This meeting is not intended to be therapeutic or interventional.

Week 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, & 21 (Weekly Teams or Phone visit 12 week ActiveHeal EST (Engage-Sustain-Triumph) Program) Twelve Individualized ActiveHeal EST (Engage-Sustain-Triumph) Sessions (Group A only): Each participant in the experiment group will receive 12 occupational therapy Teams or phone calls. This session will focus on the activities that the participants selected at the start of the program. Using the methods covered in group sessions with individualized occupational therapy intervention added. All interventions will focus on building History, Experience, Benefits, and Adaptation to optimize activity performance. More focus may be given to any of the four, based on a participant's strengths and weaknesses, at the discretion of treating therapist. All four factors must be addressed and documented per visit, and justification will be provided if a factor is not addressed (for example when a participant does not show difficulty in that domain).

Week 17 (Week 9 of active study period) Control Group B Meeting via Zoom - this study meeting lasts 15 to 30 minutes allowing the PI to touch base with the control participants to see how they are doing. This meeting is not intended to be therapeutic or interventional.

Week 22-23 Posttests - (Re-administer Occupational Resilience Measure (ORM 1.0), World Health Organization Quality of Life Scale (WHOQOL BREF), and Psychological Wellbeing Scale. To be completed with participant via Zoom. (Both Groups A & B). Group A will additionally complete Acceptability of Intervention Measure (AIM) and Feasibility of Intervention Measure (FIM).

ELIGIBILITY:
Inclusion Criteria

* Must be an adult, diagnosed within the last 12 months with prostate or breast cancer and have had treatment(s) that may be ongoing or completed.
* Must be 18-75 years old.
* Must score 80 to 90 on the Karnofsky Performance Status Scale (KPSS) Exclusion Criteria
* Unable to use or lacking access to Teams (internet) and telephone during the study period.
* Unable or unwilling to participate in activity-based interventions.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Occupational Resilience Measure (ORM 1.0) | Week 7-8; Week 22-23
  The ability to persist in selected daily activity despite challenges

SECONDARY OUTCOMES:
World Health Organization Quality of Life Scale (WHOQOL-BREF) | Week 7-8; Week 22-23
  Overall quality of life
Psychological Wellbeing Scale | Week 7-8; Week 22-23
  Wellbeing

OTHER OUTCOMES:
Acceptability of Intervention Measure- Experiment Group only | Week 22-23
  Survey
Feasibility of Intervention Measure- Experiment Group only | Week 22-23
  Survey

CONTACTS AND LOCATIONS:
Locations (1):
- University of Arkansas for Medical Science, Fayetteville, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No